CLINICAL TRIAL: NCT00829543
Title: Guide-Free Sacroiliac Injection in Spondyloarthropathies
Brief Title: Unguided Sacroiliac Injection: Effect on Refractory Buttock Pain in Patients With Spondyloarthropathies
Status: Unknown | Phase: Early Phase 1 | Type: Interventional
Last Known Status: Enrolling by invitation
Sponsor: Tabriz University (Other)
Responsible Party: Dr Shahram Sadreddini, Assistant professor of Rheumatology, Tabriz university (medical sciences)
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 8715
Record Dates: First submitted 2009-01-26; First posted 2009-01-27 (Estimated); Last update posted 2009-02-03 (Estimated); Status verified 2009-02

CONDITIONS: Spondylarthropathy
Keywords: Spodyloarthropathy; Guide-free sacroiliac injection
MeSH Terms: conditions — Spondylarthropathies

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- sacroiliac injection (Experimental): an open label study designed to evaluate the efficacy and safety of guide-free sacroiliac injection in refractory sacroiliac pain due to spondyloarthropathies
  Interventions: Procedure: guide-free sacroiliac corticosteroid injection

INTERVENTIONS:
Procedure: guide-free sacroiliac corticosteroid injection — guide-free sacroiliac injection of triamcinolone acetonide 40 mg in each sacroiliac joint
  Other Names: Unguided sacroiliac injection

SUMMARY:
This study is designed to evaluate the efficacy and safety of guide-free sacroiliac joint (SIJ) injection in refractory sacroiliac pain due to spondyloarthropathies.

DETAILED DESCRIPTION:
A 20 weeks open-label clinical trial study of 35 patients, with different subtypes of spondyloarthropathies, is conducted In spondyloarthropathy's patients with refractory inflammatory buttock pain (fulfilling inclusion criteria), we performed outpatient guide-free sacroiliac injection of triamcinolone acetonide 40 mg in each joint. Patient (pain, stiffness, sleep disturbance) and Clinician assessments (sacroiliac tenderness, Finger to floor and Schober tests ) are recorded at baseline and every 4 weeks until the end of the study. MRI scoring of sacroiliac joint is recorded according to the Spondyloarthritis Research Consortium of Canada (SPARCC) magnetic resonance imaging (MRI) index for scoring inflammatory lesions in the sacroiliac joints, at baseline and in the end of the study.

ELIGIBILITY:
Inclusion Criteria:

Patients had to fulfill the European Spondylarthropathy Study Group criteria for SpA.

1. The presence of inflammatory buttock pain for at least 4 months (typical night pain and morning stiffness) despite of receiving NSAIDs, corticosteroid and DMARDs (Disease Modifying Anti-Rheumatic Drugs) such as: methotrexate, sulfasalazin and azathioprine.
2. Tenderness over sacroiliac joint: pain over the sacroiliac sulcus with 4-5 kg/cm2 direct pressure.

Exclusion Criteria:

1. Spinal infections (such as Brucellosis).
2. Local infection in the site of injection.
3. Sacroiliac ankylosis based on pelvic X-Ray (sacroilitis grade IV).
4. Patients who had received anti TNF, corticosteroid pulse or an investigational drugs during 4 months before.

Ages: 16 Years to 50 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 35 (Estimated)
Dates: Start 2004-09; Primary Completion 2007-01 (Actual); Study Completion 2009-02 (Estimated)

PRIMARY OUTCOMES:
Refractory inflammatory sacroiliac pain | 8 months

SECONDARY OUTCOMES:
ESR, CRP | 8 months
Patient's assessment of: pain, sleep disturbance, morning stiffness | 8 months
Clinician assessment of: SIJ pain, change of finger to floor (cm) and Schober tests (mm) | 8 months
MRI SIJ inflammatory scoring | 8 months

CONTACTS AND LOCATIONS:
Overall Officials: Shahram Sadreddini, Rheumatology, Study Director — Tabriz medical university (Rheumatology Department); Shahram Sadreddini, Rheumatology, Study Chair — Assistant professor of Tabriz medical university; Mahshid Molaeefard, MD, Principal Investigator — Tehran medical university; Seyed-Kazem Shakouri, Physiatrist, Principal Investigator — Assistant professor of Tabriz medical university; Morteza Ghojazadeh, Physiologist, Principal Investigator — Assistant professor of Tabriz medical university; Hamid Noshad, Nephrologist, Principal Investigator — Assistant professor of Tabriz medical university; Mohammad-Reza Ardalan, Nephrologist, Principal Investigator — Assistant professor of Tabriz medical university
Locations (1):
- Tabriz Medical University, Rheumatology Department, Tabriz, East Azarbayjan, Iran